CLINICAL TRIAL: NCT06572956
Title: Clinical Study on the Safety and Efficacy of CAR-T/CAR-NK Cells in the Treatment of Recurrent Refractory or Unresectable Solid Tumors
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024 car-t/nk solid tumors
Record Dates: First submitted 2024-08-13; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Safety and Efficacy of Cellular Drugs, Objective Response Rate of Subjects, Etc

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- recurrent or unresectable solid tumors (Experimental): One to two days after completion of eluvial chemotherapy, CAR-T/CAR-NK cells were transfused in subjects assessed by the investigators as eligible for infusion. The CAR-T/CAR-NK dose is calculated according to the patient's body weight, and the total number of cells transfused is about 1-2x106 /kg. Single intravenous infusion.
  Interventions: Biological: CAR-T/CAR-NK cell injection

INTERVENTIONS:
Biological: CAR-T/CAR-NK cell injection — One to two days after completion of eluvial chemotherapy, CAR-T/CAR-NK cells were transfused in subjects assessed by the investigators as eligible for infusion. The CAR-T/CAR-NK dose is calculated according to the patient's body weight, and the total number of cells transfused is about 1-2x106 /kg. Single intravenous infusion.

SUMMARY:
To investigate the safety and efficacy of CAR-T/CAR-NK cells in patients with recurrent or unresectable solid tumors, including pancreatic cancer, prostate cancer, breast cancer, glioma, etc

DETAILED DESCRIPTION:
To investigate the safety and efficacy of CAR-T/CAR-NK cells in patients with recurrent or unresectable solid tumors, including pancreatic cancer, prostate cancer, breast cancer, glioma, etc.

The study was divided into five stages: screening period, single harvest period, pretreatment chemotherapy period, treatment period, observation and follow-up period after treatment.

Subjects were pretreated with FC regimen before transfusion, and the subjects who met the infusion conditions were given CAR-T/CAR-NK cell infusion 1 ~ 2 days after the completion of eluent chemotherapy. The CAR-T/CAR-NK dose is calculated according to the patient's body weight, and the total number of cells transfused is about 1-2x106 /kg. Single intravenous infusion.

The efficacy was evaluated according to the evaluation criteria for solid tumors (RECIST1.1 selection).

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent or unresectable solid tumors (including pancreatic, prostate, breast, glioma, etc.).
2. Age over 15 and under 80.
3. KPS≥50 or ECOG score ≤2 and expected survival greater than 3 months.
4. No systemic therapy (except systemic immune checkpoint suppression or activation therapy) for at least 2 weeks or at least 5 drug half-lives (whichever is shorter) prior to apheresis.
5. The absolute number of neutrophils was > 1.0x109 /L.
6. Absolute number of platelets > 50x109 /L.
7. Absolute number of lymphocytes ≥ 0.2x109 /L.
8. ALT/AST < 3 times normal value.
9. Total bilirubin < 1.5mg/dl.
10. Creatinine < 2.5mg/dl, or creatinine clearance ≥60 mL/min/1.73 m2.
11. The ejection fraction of heart ≥ 45%, echocardiography examination centerless fluid, electrocardiogram normal
12. Blood oxygen saturation ≥92% under normal environment.
13. Women of childbearing age who had a negative urine pregnancy test before dosing began and agreed to take effective contraception during the trial until the last follow-up visit.
14. Volunteer to participate in this experiment and sign the informed consent.

Exclusion Criteria:

* 1) Those who are expected to survive less than 3 months. 2) Patients whose disease progression was so rapid that a complete treatment cycle could not be ensured at the time of enrollment as determined by the investigator.

  3) Patients with primary tumors other than melanoma skin cancer (unless cured for more than 3 years).

  4) Patients with infections including fungal, bacterial, viral or other uncontrolled infections or those requiring level 4 isolation.

  5) HIV, HBV, HCV positive patients. 6) Patients with central nervous system diseases including stroke, epilepsy, dementia or autoimmune central nervous system diseases.

  7) Myocardial infection, cardiac angiography or stenting, active angina pectoris or other significant clinical symptoms, or cardiogenic asthma or cardiovascular plasma cell infiltration in the 12 months prior to enrollment.

  8) Those who are receiving anticoagulation therapy or have severe coagulation dysfunction.

  9) The drug treatment that the patient is receiving will affect the safety and efficacy study of this project according to the judgment of the investigator.

  10) Patients with allergy or history of allergy to the biologics used in this project.

  11) Pregnant or lactating women. 12) Systematic use of systemic or systemic steroid drugs within 2 weeks prior to treatment (except those who have recently or currently used inhaled steroids).

  13) The efficiency of T cell transduction by replication-deficient lentivirus was less than 30%, or the ability to expand in response to CD3 / CD28 costimulatory signals was insufficient (<5 times).

  14) Those who have other uncontrolled diseases that the researchers consider unsuitable for enrollment.

  15) Any situation that the investigator believes may increase the risk to the subject or interfere with the test results.

  16) Patients who are also participating in other clinical studies.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 2024.11
  Proportion of patients with PR or CR.
PFS | 2024.11
  The time from the start of a randomized clinical trial until tumorigenesis (any aspect) progresses or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Province, Jinan, Shandong, China